CLINICAL TRIAL: NCT04747249
Title: Psychological Care of Oncology Patients With Post-traumatic Stress in the Context of a COVID-19
Acronym: COVIPACT 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-A03234-35
Record Dates: First submitted 2021-02-08; First posted 2021-02-10 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Solid Carcinoma; Post Traumatic Stress Disorder; Covid19
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; COVID-19

STUDY DESIGN:
Intervention Model Description: Psychological support
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychological support (Experimental): Monthly psychological support
  Interventions: Other: Psychological support

INTERVENTIONS:
Other: Psychological support — Psychological care will be based on a monthly interview lasting approximately 45 minutes for 6 months.

SUMMARY:
In the context of the COVID-19 pandemic, concerns of the risk of infection may lead to fear, anxiety or psychological disorders that may become generalised and long-lasting, corresponding to post-traumatic stress disorder (PTSD). PTSD generally occurs in circumstances such as terrorist attacks, hostage-taking, bombings, aggression, accidents... The current health crisis also represents an increased risk of PTSD.

After the first moments of stress, the illness becomes more diffuse: personality change (introverted/extraverted), sleep disorders, heart problems, hypervigilance reaction, agoraphobia, symptoms of reminiscence, irritability, decreased concentration, memory loss... In some people, PTSD can lead to more disabling problems such as (crowd) avoidance.

In order to help patients with PTSD, clinical psychology offers therapeutic approaches which, starting from a debriefing with the patient, provide supportive therapy which (i) reassures by providing information on the symptomatology, in order to play down the present state of mind, (ii) allows for the expression of what was experienced during the event, (iii) initiates a process of elaboration of the trauma through transference.

A study initiated at the François Baclesse Centre during the first confinement, which included 735 patients from April to June 2020, made it possible to assess the impact of the pandemic linked to COVID-19 on the care of cancer patients treated in day hospitals, but also to evaluate the PTSD experienced by patients, sleep difficulties, quality of life, cognitive complaints and confinement conditions using validated questionnaires. This study showed that 21% of patients had proven PTSD and 23% had insomnia problem.

This study proposes to evaluate the value of adapted psychological care for patients with PTSD in relation to the pandemic on the improvement of PTSD, as well as on resilience, quality of life and sleep.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* Patient treated or followed up for a solid tumour at the François Baclesse Centre
* Patient with a score suggesting moderate or high posttraumatic stress symptoms (IES-R score ≥ 24) related to the COVID-19 epidemic
* The patient's state of health is compatible with the programme: psychological care for 6 months.
* Information note signed by the patient
* Any associated geographical, social or psychopathological conditions that might compromise the patient's ability to participate in the study

Exclusion Criteria:

* Patient with no symptoms suggestive of moderate or high post-traumatic stress (IES-R score <24)
* Patient deprived of liberty or under guardianship
* Patient already receiving psychological care
* Patient whose diagnosis of the disease was made within one month prior to the proposal for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with improvement in post-traumatic stress symptoms | 6 months

SECONDARY OUTCOMES:
Resilience Scores | 6 months
  Done with Connor-Davidson Resiliency Scale

CONTACTS AND LOCATIONS:
Overall Officials: Antony NARAYANASSAMY, M, Principal Investigator — Centre François Baclesse
Locations (1):
- Centre Francois Baclesse, Caen, France

IPD SHARING:
Plan to Share IPD: No